CLINICAL TRIAL: NCT04055766
Title: DeepDoc - Clinical Validation of an AI-based Decision Support System in the Early Diagnostic Evaluation of Neurological Diseases: a Prospective Multi-center Study
Brief Title: A Diagnostic Test on DeepDoc-an AI-based Decision Support System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DeepDoc-M5
Record Dates: First submitted 2019-08-04; First posted 2019-08-14 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-07

CONDITIONS: Stroke; Headache; Vertigo; Meningitis/Encephalitis
Keywords: Artificial Intelligence
MeSH Terms: conditions — Stroke; Headache; Vertigo; Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Meningitis/Encephalitis: Patients with clinical signs and symptoms suspected of meningitis/encephalitis
  Interventions: Device: DeepDoc AI-based Decision Support System
- Stroke: Patients with clinical signs and symptoms suspected of stroke
  Interventions: Device: DeepDoc AI-based Decision Support System
- Headache: Patients with clinical signs and symptoms suspected of headache
  Interventions: Device: DeepDoc AI-based Decision Support System
- Vertigo: Patients with clinical signs and symptoms suspected of vertigo
  Interventions: Device: DeepDoc AI-based Decision Support System

INTERVENTIONS:
Device: DeepDoc AI-based Decision Support System — Patients are diagnosed by the DeepDoc within 24 hours of admission.

SUMMARY:
DeepDoc is an AI-based decision support system for the early etiology diagnosis of neurological diseases using clinical data points from patients admitted to hospital within 24 hours.This study aims to evaluate whether the diagnosis of the DeepDoc AI-based decision support system is better than the doctor's initial diagnosis by a multi-center, superiority diagnostic study.

DETAILED DESCRIPTION:
The doctor completes the admission note within 24 hours after the patient is admitted to the hospital. After informed consent is given to the patient who meet the inclusion criteria, open the DeepDoc to fill in the patient identification information. Then take the picture of the initial diagnosis of the admission note page and upload it to DeepDoc, fill the doctor's initial diagnosis into the DeppDoc. And put the patient's clinical data points into the DeepDoc to get a DeepdDoc diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical symptoms or signs suspected of stroke，meningitis/encephalitis, vertigo and headache.
2. Neurological examination results and imaging changes within 24 hours of admission.

Exclusion Criteria:

Patients discharged, transferred to the hospital, or died within 24 hours after admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4000 consecutive patients suspected of stroke，meningitis/encephalitis, vertigo and headache（1000 cases of each disease) are admitted to the department of neurology that consented to involvement in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-09 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of diagnosis by DeepDoc AI-based Decision Support System | 24 hours
  Accuracy of diagnosis by DeepDoc and compare this result with doctors

SECONDARY OUTCOMES:
Sensitivity of diagnosis by DeepDoc AI-based Decision Support System | 24 hours
  Sensitivity of diagnosis by DeepDoc and compare this result with doctors
Specificity of diagnosis by DeepDoc AI-based Decision Support System | 24 hours
  Specificity of diagnosis by DeepDoc and compare this result with doctors

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Gang, Study Director — Xijing Hospital